CLINICAL TRIAL: NCT04876014
Title: A Guided Mobile-Based Perinatal Mindfulness Intervention - A Randomized Control Trial
Brief Title: A Guided Mobile-Based Perinatal Mindfulness Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Ng Siuman, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17603520
Record Dates: First submitted 2021-03-30; First posted 2021-05-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Psychological Distress; Mental Health Wellness 1
Keywords: Perinatal; Mindfulness; Intervention; Mobile-based; Randomized controlled trial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMBPMI group (Experimental): Participants in the experimental group will receive GMBPMI. A new participant (a pregnant woman in the second trimester) is expected to complete the 6 EBMI lessons in 6 weeks, and do the mindfulness practice for about 30-60 minutes daily. The project RA will send prompt and guidance for daily mindfulness practice to each participant through social media platform. Participants will also be asked to keep log of daily mindfulness practice from T0 to T3 using Google Form. The project RA will be available online to support, and will initiate chat every week throughout the whole intervention period. The chats will focus on participants' experiences or difficulties of mindfulness practice. The RA is backed up by the PI and co-I's who are experienced mental health practitioner and mindfulness teacher. One of them is an obstetrics and gynaecology specialist.
  Interventions: Other: Guided Mobile-Based Perinatal Mindfulness Intervention
- Perinatal Psycho-education group (Active Comparator): To control for attention and placebo effects, every new participant in the control group will receive weekly web-based psychoeducation program for perinatal care. The project RA will also be available online to support, and will initiate chat every week throughout the whole intervention period. The chats will focus on participants' experiences of the psychoeducation program.
  Interventions: Other: Guided Mobile-Based Perinatal Mindfulness Intervention

INTERVENTIONS:
Other: Guided Mobile-Based Perinatal Mindfulness Intervention — GMBPMI includes 6 EBMI lessons in 6 weeks, and it will require the participants to do mindfulness practice for about 30-60 minutes daily. The project RA will send prompt and guidance for daily mindfulness practice to each participant through social media platform. The RA will be available online to support, and will initiate chat every week throughout the whole intervention period. The chats will focus on participants' experiences or difficulties of mindfulness practice.
  Other Names: GMBPMI

SUMMARY:
Psychological distress commonly occurs among women during perinatal period. maternal psychological distress can also bring negative influence on neonatal outcomes, such as infant health, child development or mother-child interaction. Hence, developing interventions to improve mental wellbeing during this period is vital. Mindfulness based intervention (MBI) was found effective in reducing psychological distress. Most currently, delivering MBIs via internet, which is more accessible and inexpensive, shows promising positive effect in reducing psychological distress. However, randomized control trial with sufficient power is await to further confirm the positive effect among pregnant women. Moreover, the positive effects of MBIs was found associated with the heart rate variability biofeedback. However, the efficacy of MBI on HRV is rarely studied among pregnant women. Also, the potential association of HRV between MBI and psychological wellbeing needs further examination. This research aims to test the effectiveness of the Guided-Mobile Based Perinatal Mindfulness Intervention (GMBPMI) among pregnant women experiencing psychological distress during the pre and post-natal period, as well as examining the efficacy of GMBPMI on HRV.

DETAILED DESCRIPTION:
BACKGROUND Being pregnant, giving birth and turning into a mother are three closely intertwined major life transitions that a woman would experience within a short period of time. This period is often clouded by intense distress due to dramatic physical and psychosocial changes. In Hong Kong, a highly competitive and work-intense society, women face pressures on all fronts. Hong Kong ranks among the fifth with the oldest first-time mother in the world. Pregnancy at an older age is a known risk factor for antenatal depression. Women's labor force participation rate in Hong Kong is high - 84.1% in the 20-39 age group. The difficulty of balancing work and life is amplified when a woman is pregnant.

The adverse consequences of stress are broad and far-reaching, shaping obstetric and neonatal outcomes, including increased analgesic use and unplanned cesarean delivery, preterm delivery, low birth weight and Apgar scores, smaller head circumference and major congenital anomalies. Research started to reveal that the disrupting maternal cardiovascular system in pregnant women with elevated psychological distress, indexed by low heart rate variability (HRV), might be a mechanism for the worsening of birth outcomes. However, the finding is not conclusive.

In the recent decade, empirical research supporting the efficacy of prenatal mindfulness-based interventions (MBI) has emerged. MBI cultivates abilities that are important to pregnant women and new mothers, such as savoring, self-acceptance and psychological flexibility. In Hong Kong, the investigators developed and evaluated a cultural-sensitive MBI - Eastern-Based Meditation Intervention (EBMI) for pregnant women. The intervention not only showed significantly positive effects on prenatal distress coping and salivary cortisol reduction, but also associated with positive infant outcomes, including a higher cord blood cortisol level at birth and a less difficult temperament. Higher cord blood cortisol levels are believed to protect against the development of neonatal health abnormalities.

While the efficacy of prenatal MBI has been revealed in the past decade, the availability and usage of the programme remain low for various practical reasons. Moreover, providing only a limited number of lessons, mostly in the second trimester, seems insufficient. It is highly desirable to provide extended support so as to ensure continued mindfulness practice in both pre and postnatal period.

Considering the predicaments of pregnant woman/new mother, a guided mobile-based MBI appears to be more feasible than the traditional face-to-face mode. Grounded on EBMI, the investigators developed and satisfactorily piloted a guided mobile-based perinatal mindfulness intervention (GMBPMI).

OBJECTIVE and DESIGN The project aims to rigorously evaluate GMBPMI. The research adopts a parallel-armed, randomized controlled trial design. To control for confounding effects, such as attention and placebo effect, the trial will utilize an active control group. Participants in the control group will receive psychoeducation on perinatal care mimic the schedule and level of support of the experimental group.The target sample size is 198.

Pregnant women in the second trimester will be recruited to the program. With the support of a trained research assistant (RA), participants can take the 6 weekly EBMI lessons online flexibly at home. The RA will provide continued prompt and support for mindfulness practice to each participant till 5 weeks postpartum. The RA is backed up by the PI and co-I's who are experienced mental health practitioners and mindfulness teachers. One of them is an experienced obstetrics and gynaecology specialist.

EXPECTED OUTCOME In Hong Kong, around 50,000 newborn babies are delivered each year. To meet the service needs of this scale, it is imperative for us to develop a cost-effective, accessible and acceptable intervention, tailored to the predicaments of women during the perinatal period. To address the barrier and cost issues, a guided mobile-based perinatal mindfulness intervention appears to be a good choice. If the model is shown to be effective, it can be a practical solution to a large scale mental health issue - benefiting women significantly during pregnancy, as well as enhancing the subsequent mental health outcomes of these women and the well-being of their babies.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 or above
* Pregnant Chinese women in their 2nd trimester

Exclusion Criteria:

* Not able to understand Chinese (the intervention will be delivered in Chinese)
* High-risk pregnancy status (e.g., preterm labor, placental abnormality, multiple gestations, required bed rest, or morbid obesity)
* Current psychiatric disorders that necessitated priority attention (e.g., schizoaffective disorder, bipolar disorder, or current psychosis; organic mental disorder or pervasive developmental delay; current substance abuse or dependence; imminent suicide or homicide risk)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 198 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal psychological stress-General Stress ('change' is being assessed) | Change from baseline General Stress at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  General stress will be measured by Perceived Stress Scale -10. The minimum and maximum values for each item is 1 to 4 with lower score represents lower stress.
Maternal psychological stress-Pregnancy specific stress('change' is being assessed) | Change from baseline Pregnancy specific stress at post intervention (8 weeks) and 36-week gestation.
  Pregnancy specific stress will be measured by Prenatal Distress Questionnaire-12. The minimum and maximum values for each item is 0 to 4, with lower score represents lower stress.
Maternal psychological stress-Depression('change' is being assessed) | Change from baseline Depression at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  Depression is measured by Edinburgh Postnatal Depression Scale-Chinese-10. The minimum and maximum values are 1 to 4, with higher score represents higher depressive symptoms.
Mindfulness-State mindfulness('change' is being assessed) | Change from baseline State MIndfulness at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  State mindfulness is measured bu Short-form Five Facet Mindfulness Questionnaire-Chinese-20 items. The minimum and maximum values are 0 to 4, with higher score represents higher state of mindfulness.
Mindfulness-Daily mindfulness('change' is being assessed) | Weekly changes from baseline Daily Mindfulness at 5-week postpartum.
  Daily mindfulness is measured by Daily Mindful Responding Scale - 4 items. The minimum and maximum values are 0 to 10, with higher score represents higher state of mindfulness.
Positive appraisal-Coping('change' is being assessed) | Change from baseline Coping at post intervention (8 weeks) and 36-week gestation.
  Coping is measured by Prenatal Coping Inventory - 22 items. The minimum and maximum values are 0 to 4, with higher score represents higher coping frequency.
Heart rate variability('change' is being assessed) | Change from baseline HRV at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  HRV score, with higher score represents higher physical and mental condition for the day.

SECONDARY OUTCOMES:
Psychological Well-being- Anxiety('change' is being assessed) | Change from baseline Anxiety at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  Anxiety is measured by Short-form State subscale of the State-Trait Anxiety Inventory - 6 items. The minimum and maximum values range from 0 to 4, with higher score represents higher anxiety level.
Psychological Well-being- Affect('change' is being assessed) | Change from baseline Affect at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  Affect is measured by Positive & Negative Affect Subscales of Body-Mind-Spirit Well-being Inventory 9 and 10 items. The minimum and maximum values range from 0 to 10, with higher score represents higher higher frequency of experiencing particular affect.
Psychological Well-being- Spirituality('change' is being assessed) | Change from baseline Spirituality at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  Spirituality is measured by Chinese Daily Spiritual Experience Sacle - 16 items. The minimum and maximum values range from 0 to 5, with higher score represents higher frequency of experiencing spirituality.
Physical well-being-Stagnation('change' is being assessed) | Change from baseline Stagnation at post intervention (8 weeks), 36-week gestation and 5-week postpartum.
  Stagnation is measured by Stagnation Scale - 16 items. The minimum and maximum values range from 0 to 10, with higher score represents higher stagnation level.

OTHER OUTCOMES:
Clinical outcomes-Obstetric outcomes | 5 weeks postpartum
  Obstetric outcomes includes a list of 6 questions collecting information about participant's gestational age at birth, pregnancy complications, mode of birth. They are fact data without scoring.
Clinical outcomes-Neonatal outcomes | 5 weeks postpartum
  Neonatal outcomes includes a list of 4 questions collecting information about infant's birth weight, head circumference, months of maturity, and APGAR score.They are fact information without scoring.
Individual factors-Socio-demographic | Baseline (Day 0)
  Socio-demographic includes age, gender, marital status, family income, employment, education, gestational age, parity, obstetric history, medical history, and pre-pregnancy BMI. No scoring system.
Individual factors-Social Support('change' is being assessed) | Change from baseline Social Support at post intervention (8 weeks) and 36-week gestation.
  Social support is measured by Prenatal Social Support - 4 items. The minimum and maximum values range from 1 to 4, with higher score represents higher level of social support the participant has experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Siuman Ng, PhD, Principal Investigator — HKU
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The IPD is considered to share upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available upon the completion of the research program and will be available for 5 years.
Access Criteria: The IPD is considered to share upon formal request to the corresponding authors.

REFERENCES:
- [Background] Alder J, Fink N, Bitzer J, Hosli I, Holzgreve W. Depression and anxiety during pregnancy: a risk factor for obstetric, fetal and neonatal outcome? A critical review of the literature. J Matern Fetal Neonatal Med. 2007 Mar;20(3):189-209. doi: 10.1080/14767050701209560. PMID 17437220
- [Background] Female age-related fertility decline. Committee Opinion No. 589. Obstet Gynecol. 2014 Mar;123(3):719-721. doi: 10.1097/01.AOG.0000444440.96486.61. PMID 24553169
- [Background] Alderdice F, Lynn F. Factor structure of the Prenatal Distress Questionnaire. Midwifery. 2011 Aug;27(4):553-9. doi: 10.1016/j.midw.2010.05.003. Epub 2010 Sep 15. PMID 20832921
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Carlson LE, Speca M, Faris P, Patel KD. One year pre-post intervention follow-up of psychological, immune, endocrine and blood pressure outcomes of mindfulness-based stress reduction (MBSR) in breast and prostate cancer outpatients. Brain Behav Immun. 2007 Nov;21(8):1038-49. doi: 10.1016/j.bbi.2007.04.002. Epub 2007 May 22. PMID 17521871
- [Background] Bonacquisti A, Cohen MJ, Schiller CE. Acceptance and commitment therapy for perinatal mood and anxiety disorders: development of an inpatient group intervention. Arch Womens Ment Health. 2017 Oct;20(5):645-654. doi: 10.1007/s00737-017-0735-8. Epub 2017 Jun 10. PMID 28600645
- [Background] Boyd, N. G., Lewin, J. E., & Sager, J. K. (2009). A model of stress and coping and their influence on individual and organizational outcomes. Journal of Vocational Behavior, 75(2), 197-211.
- [Background] Braeken MA, Jones A, Otte RA, Nyklicek I, Van den Bergh BR. Potential benefits of mindfulness during pregnancy on maternal autonomic nervous system function and infant development. Psychophysiology. 2017 Feb;54(2):279-288. doi: 10.1111/psyp.12782. Epub 2016 Nov 7. PMID 28118687
- [Background] Byatt N, Biebel K, Friedman L, Debordes-Jackson G, Ziedonis D, Pbert L. Patient's views on depression care in obstetric settings: how do they compare to the views of perinatal health care professionals? Gen Hosp Psychiatry. 2013 Nov-Dec;35(6):598-604. doi: 10.1016/j.genhosppsych.2013.07.011. Epub 2013 Aug 19. PMID 23969144
- [Background] Chan KP. Prenatal meditation influences infant behaviors. Infant Behav Dev. 2014 Nov;37(4):556-61. doi: 10.1016/j.infbeh.2014.06.011. Epub 2014 Jul 24. PMID 25063985
- [Background] Chan, K. P. (2015). Effects of perinatal meditation on pregnant Chinese women in Hong Kong: a randomized controlled trial. Journal of Nursing Education and Practice, 5(1), 1.
- [Background] Chan, K. P. (2016). Perceptions and experiences of pregnant Chinese women in Hong Kong on prenatal meditation: A qualitative study. Journal of Nursing Education and Practice, 6(3), 135.
- [Background] Dewe, P., & Cooper, C. L. (2007). Coping research and measurement in the context of work related stress. International review of industrial and organizational psychology, 22, 141.
- [Background] Carver CS, Connor-Smith J. Personality and coping. Annu Rev Psychol. 2010;61:679-704. doi: 10.1146/annurev.psych.093008.100352. PMID 19572784
- [Background] Collins NL, Dunkel-Schetter C, Lobel M, Scrimshaw SC. Social support in pregnancy: psychosocial correlates of birth outcomes and postpartum depression. J Pers Soc Psychol. 1993 Dec;65(6):1243-58. doi: 10.1037//0022-3514.65.6.1243. PMID 8295121
- [Background] Dunkel Schetter C. Psychological science on pregnancy: stress processes, biopsychosocial models, and emerging research issues. Annu Rev Psychol. 2011;62:531-58. doi: 10.1146/annurev.psych.031809.130727. PMID 21126184
- [Background] Ecklund-Flores L, Myers MM, Monk C, Perez A, Odendaal HJ, Fifer WP. Maternal depression during pregnancy is associated with increased birth weight in term infants. Dev Psychobiol. 2017 Apr;59(3):314-323. doi: 10.1002/dev.21496. PMID 28323349
- [Background] Field T, Diego M, Hernandez-Reif M. Prenatal depression effects on the fetus and newborn: a review. Infant Behav Dev. 2006 Jul;29(3):445-55. doi: 10.1016/j.infbeh.2006.03.003. Epub 2006 May 30. PMID 17138297
- [Background] Folkman S. The case for positive emotions in the stress process. Anxiety Stress Coping. 2008 Jan;21(1):3-14. doi: 10.1080/10615800701740457. PMID 18027121
- [Background] Goodman WB, Crouter AC; The Family Life Project Key Investigators. Longitudinal Associations between Maternal Work Stress, Negative Work-Family Spillover, and Depressive Symptoms. Fam Relat. 2009 Jul 1;58(3):245-258. doi: 10.1111/j.1741-3729.2009.00550.x. PMID 20161088
- [Background] Goodman JH, Tyer-Viola L. Detection, treatment, and referral of perinatal depression and anxiety by obstetrical providers. J Womens Health (Larchmt). 2010 Mar;19(3):477-90. doi: 10.1089/jwh.2008.1352. PMID 20156110
- [Background] Guardino CM, Schetter CD. Coping during pregnancy: a systematic review and recommendations. Health Psychol Rev. 2014;8(1):70-94. doi: 10.1080/17437199.2012.752659. Epub 2014 Jan 8. PMID 24489596
- [Background] Halbreich U. The association between pregnancy processes, preterm delivery, low birth weight, and postpartum depressions--the need for interdisciplinary integration. Am J Obstet Gynecol. 2005 Oct;193(4):1312-22. doi: 10.1016/j.ajog.2005.02.103. PMID 16202720
- [Background] Hong Kong Census and Statistics Department. (2019, Aug 15). Hong Kong Monthly Digest of Statistics. Retrieved from: https://www.statistics.gov.hk/pub/B10100022018MM09B0100.pdf
- [Background] Howard LM, Piot P, Stein A. No health without perinatal mental health. Lancet. 2014 Nov 15;384(9956):1723-4. doi: 10.1016/S0140-6736(14)62040-7. Epub 2014 Nov 14. No abstract available. PMID 25455235
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Hughes A, Williams M, Bardacke N, Duncan LG, Dimidjian S, Goodman SH. Mindfulness approaches to childbirth and parenting. Br J Midwifery. 2009 Oct 1;17(10):630-635. doi: 10.12968/bjom.2009.17.10.44470. PMID 24307764
- [Background] Isgut M, Smith AK, Reimann ES, Kucuk O, Ryan J. The impact of psychological distress during pregnancy on the developing fetus: biological mechanisms and the potential benefits of mindfulness interventions. J Perinat Med. 2017 Dec 20;45(9):999-1011. doi: 10.1515/jpm-2016-0189. PMID 28141546
- [Background] Kingston D, Austin MP, Heaman M, McDonald S, Lasiuk G, Sword W, Giallo R, Hegadoren K, Vermeyden L, van Zanten SV, Kingston J, Jarema K, Biringer A. Barriers and facilitators of mental health screening in pregnancy. J Affect Disord. 2015 Nov 1;186:350-7. doi: 10.1016/j.jad.2015.06.029. Epub 2015 Jul 29. PMID 26281038
- [Background] Lacaille, J., Sadikaj, G., Nishioka, M., Flanders, J., & Knäuper, B. (2015). Measuring mindful responding in daily life: Validation of the Daily Mindful Responding Scale (DMRS). Mindfulness, 6(6), 1422-1436.
- [Background] Lau Y. The effect of maternal stress and health-related quality of life on birth outcomes among Macao Chinese pregnant women. J Perinat Neonatal Nurs. 2013 Jan-Mar;27(1):14-24. doi: 10.1097/JPN.0b013e31824473b9. PMID 23360937
- [Background] Lau Y, Keung DW. Correlates of depressive symptomatology during the second trimester of pregnancy among Hong Kong Chinese. Soc Sci Med. 2007 May;64(9):1802-11. doi: 10.1016/j.socscimed.2007.01.001. Epub 2007 Feb 21. PMID 17316942
- [Background] Lee DT, Ngai IS, Ng MM, Lok IH, Yip AS, Chung TK. Antenatal taboos among Chinese women in Hong Kong. Midwifery. 2009 Apr;25(2):104-13. doi: 10.1016/j.midw.2007.01.008. Epub 2007 Apr 3. PMID 17408821
- [Background] Lee DT, Yip SK, Chiu HF, Leung TY, Chan KP, Chau IO, Leung HC, Chung TK. Detecting postnatal depression in Chinese women. Validation of the Chinese version of the Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1998 May;172:433-7. doi: 10.1192/bjp.172.5.433. PMID 9747407
- [Background] Leung SS, Lee AM, Chiang VC, Lam SK, Kuen YW, Wong DF. Culturally sensitive, preventive antenatal group cognitive-behavioural therapy for Chinese women with depression. Int J Nurs Pract. 2013 Feb;19 Suppl 1:28-37. doi: 10.1111/ijn.12021. PMID 23425377
- [Background] Lo HH, Ng SM, Chan CL, Lam KF, Lau BH. The Chinese medicine construct "stagnation" in mind-body connection mediates the effects of mindfulness training on depression and anxiety. Complement Ther Med. 2013 Aug;21(4):348-57. doi: 10.1016/j.ctim.2013.05.008. Epub 2013 Jun 25. PMID 23876566
- [Background] Lobel, M., Yali, A. M., Zhu, W., DeVincent, C., & Meyer, B. (2002). Beneficial associations between optimistic disposition and emotional distress in high-risk pregnancy. Psychology and health, 17(1), 77-95.
- [Background] Marcus SM. Depression during pregnancy: rates, risks and consequences--Motherisk Update 2008. Can J Clin Pharmacol. 2009 Winter;16(1):e15-22. Epub 2009 Jan 22. PMID 19164843
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Martini J, Knappe S, Beesdo-Baum K, Lieb R, Wittchen HU. Anxiety disorders before birth and self-perceived distress during pregnancy: associations with maternal depression and obstetric, neonatal and early childhood outcomes. Early Hum Dev. 2010 May;86(5):305-10. doi: 10.1016/j.earlhumdev.2010.04.004. Epub 2010 May 23. PMID 20547016
- [Background] Ng SM. Validation of the 10-item Chinese perceived stress scale in elderly service workers: one-factor versus two-factor structure. BMC Psychol. 2013 Jun 19;1(1):9. doi: 10.1186/2050-7283-1-9. eCollection 2013. PMID 25566361
- [Background] Ng, S. M., Chan, C. L., Ho, D. Y., Wong, Y. Y., & Ho, R. T. (2006). Stagnation as a distinct clinical syndrome: comparing 'Yu'(stagnation) in traditional Chinese medicine with depression. British Journal of Social Work, 36(3), 467-484.
- [Background] Ng SM, Fong TC, Tsui EY, Au-Yeung FS, Law SK. Validation of the Chinese version of Underwood's Daily Spiritual Experience Scale--transcending cultural boundaries? Int J Behav Med. 2009;16(2):91-7. doi: 10.1007/s12529-009-9045-5. Epub 2009 Mar 17. PMID 19291413
- [Background] Ng SM, Yau JK, Chan CL, Chan CH, Ho DY. The measurement of body-mind-spirit well-being toward multidimensionality and transcultural applicability. Soc Work Health Care. 2005;41(1):33-52. doi: 10.1300/J010v41n01_03. PMID 16048855
- [Background] Nyklicek I, Truijens SEM, Spek V, Pop VJM. Mindfulness skills during pregnancy: Prospective associations with mother's mood and neonatal birth weight. J Psychosom Res. 2018 Apr;107:14-19. doi: 10.1016/j.jpsychores.2018.01.012. Epub 2018 Feb 4. PMID 29502758
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Raisanen S, Lehto SM, Nielsen HS, Gissler M, Kramer MR, Heinonen S. Risk factors for and perinatal outcomes of major depression during pregnancy: a population-based analysis during 2002-2010 in Finland. BMJ Open. 2014 Nov 14;4(11):e004883. doi: 10.1136/bmjopen-2014-004883. PMID 25398675
- [Background] Shea AK, Kamath MV, Fleming A, Streiner DL, Redmond K, Steiner M. The effect of depression on heart rate variability during pregnancy. A naturalistic study. Clin Auton Res. 2008 Aug;18(4):203-12. doi: 10.1007/s10286-008-0480-1. Epub 2008 Jun 30. PMID 18592128
- [Background] Shearer, A., Hunt, M., Chowdhury, M., & Nicol, L. (2016). Effects of a brief mindfulness meditation intervention on student stress and heart rate variability. International Journal of Stress Management, 23(2), 232.
- [Background] Siu BW, Leung SS, Ip P, Hung SF, O'Hara MW. Antenatal risk factors for postnatal depression: a prospective study of Chinese women at maternal and child health centres. BMC Psychiatry. 2012 Mar 22;12:22. doi: 10.1186/1471-244X-12-22. PMID 22436053
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Lever Taylor B, Cavanagh K, Strauss C. The Effectiveness of Mindfulness-Based Interventions in the Perinatal Period: A Systematic Review and Meta-Analysis. PLoS One. 2016 May 16;11(5):e0155720. doi: 10.1371/journal.pone.0155720. eCollection 2016. PMID 27182732
- [Background] Tsuda H, Kotani T, Sumigama S, Mano Y, Nakano T, Hua L, Kikkawa F. Relationship between the cortisol levels in umbilical cord blood and neonatal RDS/TTN in twin pregnancies. J Matern Fetal Neonatal Med. 2016;29(13):2151-6. doi: 10.3109/14767058.2015.1077510. Epub 2015 Sep 15. PMID 26371513
- [Background] Underwood LG, Teresi JA. The daily spiritual experience scale: development, theoretical description, reliability, exploratory factor analysis, and preliminary construct validity using health-related data. Ann Behav Med. 2002 Winter;24(1):22-33. doi: 10.1207/S15324796ABM2401_04. PMID 12008791
- [Background] van den Heuvel MI, Donkers FC, Winkler I, Otte RA, Van den Bergh BR. Maternal mindfulness and anxiety during pregnancy affect infants' neural responses to sounds. Soc Cogn Affect Neurosci. 2015 Mar;10(3):453-60. doi: 10.1093/scan/nsu075. Epub 2014 Jun 12. PMID 24925904
- [Background] van den Heuvel MI, Johannes MA, Henrichs J, Van den Bergh BR. Maternal mindfulness during pregnancy and infant socio-emotional development and temperament: the mediating role of maternal anxiety. Early Hum Dev. 2015 Feb;91(2):103-8. doi: 10.1016/j.earlhumdev.2014.12.003. Epub 2015 Jan 8. PMID 25577496
- [Background] Woolhouse H, Brown S, Krastev A, Perlen S, Gunn J. Seeking help for anxiety and depression after childbirth: results of the Maternal Health Study. Arch Womens Ment Health. 2009 Apr;12(2):75-83. doi: 10.1007/s00737-009-0049-6. Epub 2009 Feb 13. PMID 19214705
- [Background] Zeng Y, Cui Y, Li J. Prevalence and predictors of antenatal depressive symptoms among Chinese women in their third trimester: a cross-sectional survey. BMC Psychiatry. 2015 Apr 2;15:66. doi: 10.1186/s12888-015-0452-7. PMID 25879965
- [Background] Zhang JY, Cui YX, Zhou YQ, Li YL. Effects of mindfulness-based stress reduction on prenatal stress, anxiety and depression. Psychol Health Med. 2019 Jan;24(1):51-58. doi: 10.1080/13548506.2018.1468028. Epub 2018 Apr 26. PMID 29695175
- [Result] Ng SM, Fong TC, Wang XL, Wang YJ. Confirmatory factor analysis of the stagnation scale--a traditional Chinese medicine construct operationalized for mental health practice. Int J Behav Med. 2012 Jun;19(2):228-33. doi: 10.1007/s12529-011-9146-9. PMID 21279709
- [Derived] Ng SM, Leng LL, Chan KP, Lo HH, Yeung A, Lu S, Wang A, Li HY. Study protocol of guided mobile-based perinatal mindfulness intervention (GMBPMI) - a randomized controlled trial. PLoS One. 2022 Jul 8;17(7):e0270683. doi: 10.1371/journal.pone.0270683. eCollection 2022. PMID 35802637